CLINICAL TRIAL: NCT01080833
Title: Effect of Simulator Practice on Trainees' ERCP (Endoscopic Retrograde Cholangiopancreatography) Performance in the Early Learning Period: a Multi-center Randomized Controlled Observational Study
Brief Title: Effect of ERCP Mechanical Simulator (EMS) Practice on Endoscopic Retrograde Cholangiopancreatography (ERCP) Training
Acronym: ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Bay Institute for Research and Education (Other)
Collaborators: University of California, Davis (Other); University of California, Irvine (Other); University of Arizona (Other); Phoenix VA Health Care System (U.S. Federal Agency); University of New Mexico (Other); United States Naval Medical Center, San Diego (U.S. Federal Agency); Kaiser Permanente (Other)
Responsible Party: Joseph Leung, MD, EBIRE
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBIRE-GI-004
Record Dates: First submitted 2010-03-01; First posted 2010-03-04 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Training
Keywords: EMS; ERCP; Training; Trainees

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERCP mechanical simulator practice (Active Comparator): Trainees who are offered ERCP Mechanical Simulator (EMS) training in addition to routine training (study group)
  Interventions: Device: ERCP mechanical simulator practice
- No ERCP mechanical simulator practice (No Intervention): Trainees undergoing routine ERCP training only (control group).

INTERVENTIONS:
Device: ERCP mechanical simulator practice — Trainees will receive ERCP mechanical simulator practice in addition to routine ERCP training
  Arms: ERCP mechanical simulator practice

SUMMARY:
Trainees who are offered ERCP Mechanical Simulator (EMS) training in addition to routine training (study group) will demonstrate improved clinical outcomes compared to those undergoing routine ERCP training only (control group).

DETAILED DESCRIPTION:
Hypothesis #1: Trainees who are offered simulator training in addition to routine training (study group) will demonstrate improved clinical outcomes compared to those undergoing routine ERCP training only (control group).

Hypothesis #2: Trainees who are initially in the control arm, but receive the simulator training after the initial 30 procedures (delayed intervention) will have significantly greater improvement of clinical outcomes in the second phase of the study (steeper learning curve) compared to the initial period.

STUDY DESIGN & OUTCOMES

* Controlled randomized observational study.
* Immediate intervention (simulator training in the beginning of or just prior to the trainees' ERCP rotation) and delayed intervention (simulator training after 30 clinical procedures) will be studied
* Primary outcome: diagnostic biliary cannulation and deep biliary cannulation success rates Secondary outcomes: cannulation time, subjective competency score (5-point scale) graded by supervising physicians.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal fellows receiving ERCP training

Exclusion Criteria:

* Gastrointestinal fellows who are not receiving ERCP training

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic biliary cannulation and deep biliary cannulation success rates | 12 months
  The ability of the trainees to perform solo diagnostic biliary cannulation and deep biliary cannulation

SECONDARY OUTCOMES:
Trainer assessment | 12 months
  Subjective competency (5-point score) graded by supervising physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Leung, MD, Principal Investigator — Sacramento VA Medical Center
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Leung JW, Lee JG, Rojany M, Wilson R, Leung FW. Development of a novel ERCP mechanical simulator. Gastrointest Endosc. 2007 Jun;65(7):1056-62. doi: 10.1016/j.gie.2006.11.018. PMID 17531642